CLINICAL TRIAL: NCT06542874
Title: Safety and Efficacy of Once-weekly Subcutaneous and Once-daily Oral NNC0487-0111 in Participants With Type 2 Diabetes - a Dose Finding Study
Brief Title: A Research Study Comparing How Well Different Doses of the Medicine NNC0487-0111 Lower Blood Sugar in People With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9490-7678; U1111-1296-9708 (Other: World Health Organization (WHO)); 2023-509412-28 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Placebo subcutaneous (Placebo Comparator): Placebo for subcutaneous treatment
  Interventions: Drug: Placebo (NNC0487-0111 subcutanous)
- NNC0487-0111 subcutaneous dose 1 (Experimental): NNC0487-0111 subcutaneous dose 1 treatment
  Interventions: Drug: NNC0487-0111 subcutanous
- NNC0487-0111 subcutaneous dose 2 (Experimental): NNC0487-0111 subcutaneous dose 2 treatment
  Interventions: Drug: NNC0487-0111 subcutanous
- NNC0487-0111 subcutaneous dose 3 (Experimental): NNC0487-0111 subcutaneous dose 3 treatment
  Interventions: Drug: NNC0487-0111 subcutanous
- NNC0487-0111 subcutaneous dose 4 (Experimental): NNC0487-0111 subcutaneous dose 4 treatment
  Interventions: Drug: NNC0487-0111 subcutanous
- NNC0487-0111 subcutaneous dose 5 (Experimental): NNC0487-0111 subcutaneous dose 5 treatment
  Interventions: Drug: NNC0487-0111 subcutanous
- NNC0487-0111 subcutaneous dose 6 (Experimental): NNC0487-0111 subcutaneous dose 6 treatment
  Interventions: Drug: NNC0487-0111 subcutanous
- Placebo oral (Placebo Comparator): Placebo for oral treatment
  Interventions: Drug: Placebo (NNC0487-0111 oral)
- NNC0487-0111 oral dose 1 (Experimental): NNC0487-0111 oral dose 1 treatment
  Interventions: Drug: NNC0487-0111 oral
- NNC0487-0111 oral dose 2 (Experimental): NNC0487-0111 oral dose 2 treatment
  Interventions: Drug: NNC0487-0111 oral
- NNC0487-0111 oral dose 3 (Experimental): NNC0487-0111 oral dose 3 treatment
  Interventions: Drug: NNC0487-0111 oral

INTERVENTIONS:
Drug: NNC0487-0111 subcutanous — NNC0487-0111 administered subcutanously (under the skin)
  Arms: NNC0487-0111 subcutaneous dose 1; NNC0487-0111 subcutaneous dose 2; NNC0487-0111 subcutaneous dose 3; NNC0487-0111 subcutaneous dose 4; NNC0487-0111 subcutaneous dose 5; NNC0487-0111 subcutaneous dose 6
Drug: Placebo (NNC0487-0111 subcutanous) — NNC0487-0111 placebo administered subcutanously (under the skin)
  Arms: Placebo subcutaneous
Drug: NNC0487-0111 oral — NNC0487-0111 administered orally (in the mouth)
  Arms: NNC0487-0111 oral dose 1; NNC0487-0111 oral dose 2; NNC0487-0111 oral dose 3
Drug: Placebo (NNC0487-0111 oral) — NNC0487-0111 placebo administered orally (in the mouth)
  Arms: Placebo oral

SUMMARY:
The study will look at how well different doses of a new medicine called NNC0487-0111 help lower the blood sugar and body weight in people with type 2 diabetes. NNC0487-0111 is a new medicine which cannot be prescribed by doctors but has previously been tested in humans. Participants will either get NNC0487-0111, which is given as tablets or as injections, or placebo. Which treatment the participant get is decided by chance.The study will last for about 43 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus greater or equal to 180 days before screening.
* Stable daily dose(s) greater or equal to 90 days before screening of the following antidiabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose as judged by the investigator: metformin with or without SGLT2 inhibitor.
* HbA1c of 7.0-10.0 procent (53-86 mmol/mol) (both inclusive) as assessed by central laboratory at screening.
* Body mass index between greater or equal to 23.0 and below 50.0 kg/m^2.
* Able and willing to adhere to the protocol including wearing a continuous glucose monitoring (CGM) device provided for the study, as judged by the investigator.

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to end of treatment (week 36)
  percent point

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 36)
  percent
Change in body weight | From baseline (week 0) to end of treatment (week 36)
  kg
Change in fasting plasma glucose (FPG) | From baseline (week 0) to end of treatment (week 36)
  mmol/L
CGM: Change in time in range (TIR) 3.9-10.0 mmol/L (70-180 mg/dL) | From baseline (week 0) to end of treatment (week 36)
  percent points
Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 36)
  kg/m^2
Change in waist circumference | From baseline (week 0) to end of treatment (week 36)
  cm
Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 36)
  mmHg
Change in average 24-hour systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 36)
  mmHg
Change in high sensitivity C-Reactive Protein (hsCRP) | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in total cholesterol | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in triglycerides | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Number of adverse events | From baseline (week 0) to end of study (week 40)
  Count of events
Change in Urinary Albumin/Creatinine Ratio (UACR) | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Participant without macroalbuminuria (UACR < 300 mg/g) at baseline (week 0) developing (yes/no) new onset of macroalbuminuria (UACR ≥ 300 mg/g) | At end of treatment (week 36)
  Count of participant
Change in eGFR creatinine- and cystatin C based CKD-EPI | From baseline (week 0) to end of treatment (week 36)
  mL/min/1.73 m^2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (114):
- United States (28):
  - Southern Cal Clinical Research, Santa Ana, California
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Fleming Island Ctr for Clin Res, Fleming Island, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - South Broward Research LLC, Miramar, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Advanced Internal Medicine, PLLC, Paducah, Kentucky
  - Medstar Research Institute_Hyattsville, Hyattsville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - Arcturus Healthcare, PLC, Troy, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - AMC Community Endocrinology, Albany, New York
  - Lucas Research Inc., Morehead City, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Plains Clinical Research Center, LLC_Fargo, Fargo, North Dakota
  - Preferred Primary Care Physicians_Pittsburgh, Pittsburgh, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Clinical Research Associates, Nashville, Tennessee
  - MidState Endocrine Associates, Nashville, Tennessee
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Victorium Clinical Research, Houston, Texas
  - Synergy Groups Medical, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - Tekton Research, McKinney, Texas
  - Hillcrest Family Health Center, Waco, Texas
- Bulgaria (11):
  - Individual Practice For Specialized Outpatient Medical Care Doctor Miglena Rizova Ltd., Kyustendil
  - IPSOMC Dr. Miglena Rizova Ltd., Kyustendil
  - UMHAT "Kaspela", Depart. Endocrinology and Metab. Diseases, Plovdiv
  - UMHAT Kaspela EOOD, Endocrinology and Metabolic Diseases Clinic, Plovdiv
  - DCC Sveti Georgi EOOD, Plovdiv
  - Diagnostic-Consultative Centre "Sveti Georgi" Eood, Plovdiv
  - Medical centre Regina Life Clinic EOOD, Sofia
  - UMHAT "Aleksandrovska", Sofia
  - USHATE "Akad. Ivan Penchev" Second Clinic of Endocrinology, Sofia
  - USHATE Akad. Ivan Penchev EAD, Second Clinic of Endocrinology, Sofia
  - AIPSMC Dr. Artin Magardichyan EOOD, Varna
- Croatia (10):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Clinical Hospital Centre Rijeka_Endocrinology, Rijeka, Primorje-Gorski Kotar County
  - KBC Rijeka, Endokrinologija, Rijeka, Primorje-Gorski Kotar County
  - Opca bolnica Karlovac, Karlovac
  - Specijalna bolnica Krapinske Toplice - Endokrinologija, Krapinske Toplice
  - Specijalna Bolnica za medicinsku rehabilitaciju Krapinske Toplice_Endocrinology, Krapinske Toplice
  - Klinicki bolnicki centar Osijek_Endocrinology, Osijek
  - Klinicki bolnicki centar Osijek, Osijek
  - Opca bolnica Varazdin_Endocrinology, Varaždin
  - Opca bolnica Varazdin, Varaždin
- Germany (6):
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Wendisch/Dahl Hamburg, Hamburg
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
- Greece (7):
  - Iatriko Psychicou Private Clinic, Athens
  - U.G.H of Athens "Attikon", Athens
  - "Laiko" General Hospital of Athens, Goudi/Athens
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - 424 Military General Training Hospital - 2nd Department of Internal Medicine, Thessaloniki
  - 424 Military General Training Hospital, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
- Hungary (6):
  - Debreceni Egyetem, Debrecen, Hajdú-Bihar
  - Bajcsy-Zsilinszky Kórház, Budapest
  - MH Egészségügyi Központ, Budapest
  - Debreceni Egyetem, Debrecen
  - Békés Megyei Központi Kórház, Gyula
  - Somogy Vármegyei Kaposi Mór Oktató Kórház, Kaposvár
- Japan (12):
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Heiwadai Hospital, Miyazaki, Miyazaki
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Tokuyama clinic, Chiba
  - Akaicho Clinic, Chiba-shi, Chiba
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Naka Kinen Clinic, Ibaraki
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
- Poland (13):
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Formed 2 Sp. z o.o., Oświęcim, Lesser Poland Voivodeship
  - Beata Miklaszewicz & Dariusz Dabrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - Beata Mikłaszewicz & Dariusz Dąbrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - EKAMED sp. z o.o., Lublin, Lublin Voivodeship
  - ETG Siedlce, Siedlce, Masovian Voivodeship
  - Specderm Poznanska Sp. j., Bialystok, Podlaskie Voivodeship
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Specderm Poznańska Spółka Jawna, Bialystok
  - EKAMED sp. z o.o., Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Specjalistyczna A Wittek H Rudzki Sp. j., Ruda Śląska
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
  - Santa Sp. z o.o, Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz, Łódź Voivodeship
- Romania (8):
  - SC Grand Med SRL, Oradea, Bihor County
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Spitalul Clinic Judetean Urgenta Cluj-Napoca, Cluj-Napoca, Cluj
  - Sc Mediab Srl, Târgu Mureş, Mureș County
  - Novus Medical Clinica SRL, Ploieşti, Prahova
  - Mariodiab Clinic SRL, Brasov
  - Cabinet Medical Dr Geru SRL, Timișoara
  - Spitalul Clinic Judetean De Urgenta Pius Brinzeu Timisoara, Timișoara
- Slovakia (5):
  - Peter Farkas MD, s.r.o., Šahy, Slovak Republic
  - DENTAVIA s.r.o., Poprad
  - DIABETOL, s.r.o., Prešov
  - OLIVER - MED s.r.o., Rimavská Sobota
  - MEDIVASA, s.r.o., Diabetologicka ambulancia, Žilina
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Infanta Luisa, Seville
  - Hospital Nisa Sevilla Aljarafe, Seville
  - Hospital Vithas Sevilla, Seville

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com